CLINICAL TRIAL: NCT03038841
Title: Mobile Health Technologies for Palliative Care Patients at the Interface of In-patient to Out-patient Care: A Feasibility Study Aiming to Early Predict Deterioration of Patient's Health Status
Brief Title: Mobile Health Technology for Palliative Care Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Zurich (Other)
Collaborators: Swiss Federal Institute of Technology (Other); Swiss Academy of Medical Sciences (SAMS) (Other)
Responsible Party: Sponsor
Other Study IDs: PC 16/16
Record Dates: First submitted 2017-01-25; First posted 2017-02-01 (Estimated); Last update posted 2017-06-21 (Actual); Status verified 2017-01

CONDITIONS: Metastatic Cancer; Mobile Health; Chronic Disease
MeSH Terms: conditions — Neoplasm Metastasis; Chronic Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Mobile Health — Patients discharged from hospital will be equipped with a tracking bracelet and a smart phone

SUMMARY:
To test the potential and acceptance of wireless activity tracking in palliative care patients leaving hospital care. Explorative study, collaboration project of the Clinic of Radiation-Oncology, University Hospital Zurich and the Wearable Computing Laboratory, Swiss Federal Institut of Technology. Patients receive a tracking bracelet and a smart phone in order to gather objective physical activity parameters as step count, sleep duration, heart rate, social activity patterns (e.g. making calls) as well as subjective ratings of pain and distress. Quality of life (QoL) will be captured by paper questionnaire. Correlations between patients' physical activity patterns and the pain and distress level assessed from electronic scales as well as QoL-questionnaire will be performed. Acceptance will be evaluated by quantitative questionnaires and interviews. The proposed study is meant to be preparatory work for an intervention study to test the effect of wireless monitoring of palliative care patients on fostering early interventions for symptom relief and support of QoL.

ELIGIBILITY:
Inclusion Criteria:

* established diagnosis of metastatic cancer or other severe illness with limited life-expectancy (physicians guess <12 months, > 8 weeks)
* Karnofsky Index ≥50%
* ECOG≤ 2
* aged > 18 years
* passed a short handling test with devices (tracking bracelet, smart phone)

Exclusion Criteria:

* relevant cognitive impairment
* insufficient knowledge of German language.

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients hospitalized at one of the wards of the Clinic of Radiation-Oncology University Hospital Zurich, including a ward of specialized Palliative Care
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2018-05-31 (Estimated); Study Completion 2018-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility (time of complete data transfer in weeks) | 12 weeks
  time of complete data transfer in weeks

CONTACTS AND LOCATIONS:
Overall Officials: Matthias Guckenberger, Prof, Study Chair — Clinic of Radiation-Oncology USZ; Gerhard Tröster, Prof, Study Chair — ETH Zürich; Gudrun Theile, MD, Principal Investigator — Clinic of Radiation-Oncology USZ
Locations (1):
- Clinic of Radiation-Oncology University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No